CLINICAL TRIAL: NCT03998605
Title: Protect Yourself: Abuse Prevention for People With Intellectual Disabilities
Acronym: AP4ID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no release of remaining funds
Sponsor: Double S Instructonal Systems (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AbusePhaseII; R44HD079119-02 (NIH)
Record Dates: First submitted 2019-06-22; First posted 2019-06-26 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Abuse Prevention
Keywords: intellectual disabilities; abuse; abuse prevention
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abuse Prevention Program Condition (Experimental): The abuse prevention program will address: (1) BEFORE -- (a) Learning about problem of abuse and what abuse is; (b) Knowing about types of abuse, who the abusers are and where abuse happens; (c) Planning ahead and identifying safe people; (2) DURING -- (a) Rejecting abuse by saying "no;" (b) Getting away if possible/staying safe and paying attention, (c) Staying calm and getting home; and (3) AFTER -- (a) Telling your safe person, (b) Knowing what to do and what not to do, and (c) Reporting the abuse and getting help to cope with the event.
  Interventions: Behavioral: Abuse Prevention Program
- Control condition (Active Comparator): During the study the control group will receive 12 activity sheets from the ESCAPE-NOW curriculum. Six activity sheets will be given at the initial meeting and half way through the study the remaining activity sheets will be mailed to the dyads. We chose these activity sheets because they provide abuse information that was designed for individuals with ID.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Abuse Prevention Program — The abuse prevention program will be comprised of nine shared learning modules for the individual with Intellectual Disabilities (ID) and a care provider. Each shared module will contain an action step in the Individual Response Plan and will include video, guided practice and workbook activities to equip persons with ID with a range of judgment, decision-making skills and the efficacy needed for identifying, rejecting, and reporting abuse.
  Arms: Abuse Prevention Program Condition
Behavioral: Control Condition — The control group will receive worksheets from the ESCAPE-NOW curriculum.
  Arms: Control condition

SUMMARY:
The purpose of this study is to help individuals and their caregivers develop a plan on how to recognize, deal with and respond to abusive situations.

DETAILED DESCRIPTION:
The goal of this project is to address the current deficiencies by creating a program that will guide individuals who have intellectual disabilities and a Learning Partner (LP - care provider, relative, group home staff) in developing a comprehensive Individual Response Plan (IRP) that can be used before, during, and after an abusive event. Behavioral skills training and behavioral relaxation training -- two instructional approaches with evidence for effectiveness in this population -- will be included to address the unique learning needs of people who have intellectual disabilities and to maximize opportunities for skill-based learning. Video and workbook activities will train the LP to effectively implement the abuse prevention and response strategies, thus increasing the potential for generalization in the natural environment and long-term maintenance of skills.

ELIGIBILITY:
Inclusion Criteria:

* has moderate to mild mental retardation based on IQ scores ranging from 40-70
* is over 18 years old. --the participant must be able to do three of the following four skills (1) complete a simple worksheet with assistance, (2) go on simple errands alone, (3) recognize 10 or more words by site, (4) read a digital clock.

Exclusion Criteria:

* individuals who have experienced traumatic abuse and experiences symptoms suggestive of trauma, such as flashbacks, nightmares, and chronic anxiety and/or depression that is resistant to standard pharmacological and psychotherapy/behavior interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-04 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Abuse Protection Concept Questionnaire | Pre, post (9 weeks), and 2 month follow-up
  This questionnaire assesses change in knowledge and attitude about various types of abuse in individuals with Intellectual Disability (ID). The questionnaire includes three sub scales. The first sub-scale is comprised of five open ended questions. Score answers range from 0 to 3 with a total score of 15. Higher scores reflect higher knowledge. The second sub-scale presents structured questions about the five types of abuse. The total possible score for the first part of the second sub-scale is 5 -- with higher score reflecting greater knowledge. Participants are then shown five pictures depicting types of abuse. Each correct response was awarded a point for a total of five. The total possible score for sub-sale 2 is 10. Sub-scale 3 is a 20 item forced choice -- yes (1) , no (0), don't know (0) - that assesses knowledge and attitudes. with a total possible sub-score of 20 -- higher score equals higher knowledge.
Abuse Protection Decision Making and Task Analysis Check Sheet | Pre, post (9 weeks), and 2 month follow-up
  This checklist assesses change in knowledge required by people with ID to recognize and report abuse. It consists of five vignettes of abusive situations and two non-abusive. Each vignette has a a possible score of 10. The total possible score for all seven vignettes is 70 with higher scores reflecting greater knowledge.

SECONDARY OUTCOMES:
Glascow Social Self-Efficacy Scale | Pre, post (9 weeks), and 2 month follow-up
  Change in social self-efficacy in people with moderate to mild intellectual disabilities as measured by the 17-item self-efficacy scale. A three point response format is used to answer each question: not at all, a little bit, or a lot. Responses are scored 0,1, and 2 respectively giving a range of 0-34. Higher values represent better outcomes.
Test of Interpersonal Competence and Personal Vulnerability | Pre, post (9 weeks), and 2 month follow-up
  Change in the 20-item multiple-choice interpersonal competence and vulnerability of individuals with ID. Each question has three answers with only one best answer for each question.Scoring is from 0 to 1 with 1 being the best answer. Scores range from 0 to 20 with higher scores showing improvement in interpersonal competence and personal vulnerability.
Social Vulnerability Questionnaire | Pre, post (9 weeks), and 2 month follow-up
  Change in social vulnerability in individuals with ID as measured by 45 items that assess social vulnerability. Care provider rates individual with ID on a 4-point Likert scale (1=not true or never to 4= very true or always). Scores range from 45 to 180. Lower scores reflect improvements in social vulnerability.

OTHER OUTCOMES:
Adults with ID Consumer Satisfaction | Post (9 weeks)
  This consumer satisfaction scale for people with ID consists of 15 items and 1 open-ended question that assesses relevance and clarity of materials and program use barriers. The 15 items are rated on a three point scale -1= not at all; 2= somewhat; and 3= a lot. The total possible score was 45. Higher scores reflect greater satisfaction with the program.
Learning Partner Consumer Satisfaction | Post (9 weeks)
  This consumer satisfaction scale for the care giver (Learning Partner) consists of 31 items, and 1 open-ended question to assess usability and effectiveness of materials. The five point scale ranged from 1= strongly agree to 5= strongly disagree. The total possible score was 155 with lower scores reflecting greater satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Martin R. Sheehan, Ph.D., Principal Investigator — Research Director
Locations (1):
- Double S Instructional Systems, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent reviewer. Requestors will be required to sign a data access agreement.
URL: http://doublesinstructional.com